CLINICAL TRIAL: NCT01639365
Title: Usefulness of the SmartTouch Catheter to Assess the Areas of Myocardial Scar in Patients With Ventricular Tachycardia
Brief Title: SmartTouch Catheter in Ablation of Ventricular Tachycardia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Arcadio Garcia Alberola, Professor of Cardiology, Hospital Universitario Virgen de la Arrixaca
Other Study IDs: IIS-176
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Arrhythmias, Cardiac; Tachycardia, Ventricular; Myocardial Infarction; Cardiomyopathies
Keywords: Ventricular tachycardia; Catheter ablation; Tissue contact
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia, Ventricular; Myocardial Infarction; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The pressure exerted by the ablation catheter on the tissue has been shown to play an important role on determining the size and the potential efficacy of the ablation lesions. A direct information on the force exerted by the catheter tip obtained from the SmartTouch technology might improve the assessment of the scar areas during electroanatomical mapping in patients with ventricular tachycardia (VT) due to ischemic disease or cardiomyopathy. The objectives of the study are to compare the areas of scar (defined as a low-voltage threshold) obtained from the conventional voltage map with those obtained after the contact map information is available to the operator and to determine if the availability of the contact information allows an improvement of the electroanatomic map by correcting the points taken in no-contact areas. Twenty to 30 consecutive patients with ventricular arrhythmias due to ischemic heart disease or dilated cardiomyopathy undergoing VT ablation will be included in a prospective, one-center, non-randomized study. A voltage map of the left ventricle will be obtained using the CARTO-3 navigation system and the scar areas as well as the areas of potential interest for ablation will be delineated in the standard way and saved as the control map. The force information will be recorded by the system but will not be available to the operator until the control map is saved. Following this step the contact map will be available to the operator to be compared with the control map and further mapping and point acquisition will be allowed to correct the areas previously acquired with poor or no contact. The final map after corrections have been made will be saved as the corrected map. The ablation procedure will then be performed as usual. Both maps will be compared in a deferred way to know how are classified the areas without contact when no pressure information is available, and how many non-contact points are falsely assumed to be low-voltage or dense scar points. These comparisons will give information on how much the standard electroanatomic map can be improved when the force information is added.

DETAILED DESCRIPTION:
The usual ablation catheters do not provide direct information on the pressure applied at the contact area of the cardiac structures. However, pressure has been shown to play an important role on determining the size and the potential efficacy of the ablation lesions. The physical contact of the tip of the catheter with the tissue and the force exerted on this tissue are indirectly estimated from other parameters such as the signal voltage, the transmitted force to the other end of the catheter felt by the operator and, in a lesser extent, the circuit impedance.

A widespread technique for ablation of ventricular tachycardias (VT) in patients with cardiomyopathies or ischemic disease consists on the creation of an electroanatomic map to delineate scar areas without electric activity and to look for areas of surviving myocardium inside, at the borders or between the scars, operating as a slow conduction channel in a reentry circuit and playing an essential role in the genesis of VTs. The distinction between scar and normal tissue is predominantly based on the voltage of the unipolar or bipolar electrograms (EGM) recorded at the tip of the ablation catheter. However, the amplitude of the electrogram depends critically on the distance between the electrode and the source of the electric field, in this case the myocardial tissue. The lack of contact between the catheter and the endocardium will reduce the EGM voltage and may induce to interpret a normal EGM point as a low-voltage point, leading to an erroneous delineation of the real scar areas and eventually missing electrically active myocardial paths. Thus a good physical contact between the catheter and the tissue is a prerequisite to obtain a reliable voltage map and to correctly identify scars and areas potentially involved in the VT maintenance. A direct information on the force applied at the tip of the catheter may avoid the interpretation of areas with no-contact induced low-voltage as scars.

Hypothesis.

The hypothesis of the study is that the information on the force exerted by the catheter tip obtained from the SmartTouch technology may improve the assessment of the scar areas during electroanatomical mapping in patients with VT due to ischemic disease or cardiomyopathy.

Study objectives and endpoints.

Two are the main objectives of this study:

1. To compare the areas of scar (defined as a low-voltage threshold) obtained from the conventional voltage map with those obtained after the contact map information is available to the operator.
2. To determine if the availability of the contact information to the operator allows an improvement of the electroanatomic map by correcting the points taken in no-contact areas.

Study protocol.

1. Inclusion criteria.

   Consecutive patients with ventricular arrhythmias due to ischemic heart disease or dilated cardiomyopathy undergoing VT ablation will be included in the study.

   Exclusion criteria will be age <18 years, absence of signed informed consent or critical clinical status that precludes a detailed mapping procedure.
2. Study design and duration.

   The study is planned as a prospective, one-center, non-randomized study. As the objectives are purely descriptive no formal calculation of the sample size has been performed. Considering the inclusion criteria and the frequency of this type of studies in our unit a number of 20 to 30 patients is estimated to be included in 12 months. We believe that this number of patients is reasonable to estimate the value of the contact map to delineate scars from a clinical point of view.
3. Protocol and procedure.

   Our standard approach to ischemic VT ablation begins with the acquisition of a voltage map of the left ventricle during sinus rhythm of fixed pacing from the right ventricular apex using the CARTO-3 navigation system and a Navistar irrigated catheter. During the acquisition, points with fragmented or delayed potentials are tagged as areas of potential interest for ablation. Once the map is completed we adjust the color code of the voltage map trying to decide the areas of dense scar and to look for potential narrow paths inside or between the areas of scar. After adjusting the map in this way we proceed to the ablation, which is performed during induced VT or guided by the anatomical and electrical information in case of non-inducible or non-tolerated VTs. Pace-mapping is eventually used if a 12-lead ECG of the clinical VT is available.

   For the patients included in the study the voltage map will be acquired in the same way using the Thermo-Cool Smart Touch catheter. The force information will be recorded by the system but will not be available to the operator during the map acquisition. The completed voltage map with the areas defined as dense scar by the operator, the isthmuses found inside or between scars and the areas with fragmented or delayed potentials will be saved as the control map. Following this step the contact map will be available to the operator to be compared with the control map and further mapping and point acquisition will be allowed to correct the areas previously acquired with poor or no contact. The final map after corrections have been made will be saved as the corrected map. The ablation procedure will then be performed as usual.
4. Map analysis

   The comparison of the maps will be done in a deferred way. First, the control map and the contact map will be compared. The area without contact in the pressure map will be estimated. Each point inside this area will be classified as dense scar, low-voltage point or normal voltage point according to the properties of the point in the control map. We will determine in this way how are classified the areas without contact when no pressure information is available, and how many non-contact points are falsely assumed to be dense scar. The areas of "real" dense scar and "assumed, non-contact" dense scar will be estimated as well. This step of the analysis will give information on how many low-voltage areas of the standard electroanatomic map may not be reliable due to lack of an appropriate contact.

   The control and the corrected map will then be compared. The areas and the number of points defined as dense scar by the operator in both maps will be compared and the points changing their status as scar, low or normal voltage from the control to the corrected map will be annotated as well. Finally, the differences in the potential isthmuses depicted in both maps will be analyzed. These comparisons will give information on how much the standard electroanatomic map can be improved when the force information is added.
5. Patient consent.

   The study will be presented to the ethics committee of our centre for approval. A written, informed consent will be required to be signed by the patient before entering the study.
6. Time schedule

   The recruitment of patients will start as soon as the project is approved by Biosense Webster and by the local ethics committee. The inclusion period would be 12 months. Data analysis will be performed during the study period, making the final results available shortly after the end of the study. An additional 6 month period is expected to report and publish the results in international cardiology journals.
7. Privacy policy

All the patient's data will remain in the hospital files and will not be transmitted to any external subject. A code will be assigned to each patient in order to allow the analysis of the data in an anonymous way .

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with ventricular arrhythmias due to ischemic heart disease or dilated cardiomyopathy undergoing VT ablation

Exclusion Criteria:

* Age <18 years, absence of signed informed consent or critical clinical status that precludes a detailed mapping procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with ventricular arrhythmias due to ischemic heart disease or dilated cardiomyopathy undergoing VT ablation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the scarred areas obtained by traditional voltage mapping with those obtained using a map that includes the contact force information in patients with VT | During ablation procedure
  The size of the scars, the abnormal potentials, and the channels detected in the control map were compared with those of the final map

CONTACTS AND LOCATIONS:
Overall Officials: Arcadi Garcia-Alberola, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- University Hospital Virgen de la Arrixaca, Murcia, Murcia, Spain

REFERENCES:
- [Background] Sanchez Munoz JJ, Penafiel Verdu P, Martinez Sanchez J, Salar Alcaraz M, Valdes Chavarri M, Garcia Alberola A. Usefulness of the contact force sensing catheter to assess the areas of myocardial scar in patients with ventricular tachycardia. Rev Esp Cardiol (Engl Ed). 2015 Feb;68(2):159-60. doi: 10.1016/j.rec.2014.09.011. Epub 2014 Dec 12. No abstract available. PMID 25499952
- See also: Related Info — http://www.revespcardiol.org/en/usefulness-of-the-contact-force/articulo/90376822/